CLINICAL TRIAL: NCT00075777
Title: A Pilot Trial Of Valproic Acid In Patients With Kaposi's Sarcoma
Brief Title: Valproic Acid in Treating Patients With Kaposi's Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-038; U01CA070019 (NIH); CDR0000349348 (Other: NCI)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Sarcoma
Keywords: recurrent Kaposi sarcoma; AIDS-related Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Kaposi; AIDS-related Kaposi sarcoma | interventions — Valproic Acid

INTERVENTIONS:
Drug: valproic acid — 250 mg by mouth twice a day
  Other Names: Depakene

SUMMARY:
RATIONALE: Valproic acid may help stop the growth of Kaposi's sarcoma cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: This clinical trial is studying valproic acid in treating patients with HIV-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of valproic acid in patients with Kaposi's sarcoma.
* Determine the effects of this drug on human herpes virus 8 (KSHV) gene expression using polymerase chain reaction and immunohistochemistry in these patients.

Secondary

* Determine the effects of this drug on HIV, KSHV, and Epstein-Barr virus viral loads in the plasma and peripheral blood mononuclear cells of these patients.
* Determine clinical response in patients treated with this drug.

OUTLINE: This is an open-label, pilot, multicenter study.

Patients receive oral valproic acid twice daily on days 1-28 followed by a drug taper over 2 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed HIV-related Kaposi's sarcoma (KS)

  * Disease involving the skin and/or lymph nodes

    * No symptomatic visceral disease
    * No oral KS as the only site of disease
  * Slowly progressive or stable disease allowed

    * Slow progression defined as fewer than 5 new lesions per month
  * Must have documented HIV infection by positive ELISA, western Blot, or viral load determination
* CD4 T-cell count > 50/mm^3

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)*
* AST and ALT ≤ 3 times ULN
* Albumin > 2.5 g/dL NOTE: *Elevated total bilirubin (≤ 3.5 mg/dL) secondary to indinavir therapy allowed provided the direct bilirubin is normal

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* No prior myocardial infarction
* No evidence of cardiac ischemia

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No prior lactic acidosis > 2.0 mmoles/L
* No prior lipoatrophy or hypercholesterolemia secondary to retroviral treatment
* No concurrent, acute, active opportunistic infection other than oral thrush or genital herpes within the past 14 days
* No other concurrent neoplasm requiring cytotoxic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior biologic therapy for KS

Chemotherapy

* More than 2 weeks since prior chemotherapy for KS
* No concurrent systemic cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 2 weeks since prior radiotherapy for KS

Surgery

* Not specified

Other

* More than 2 weeks since other prior antineoplastic or local therapy for KS
* More than 2 weeks since prior investigational therapy for KS
* More than 60 days since prior local therapy to a KS-marker lesion unless lesion has clearly progressed since therapy
* More than 1 year since prior valproic acid
* Concurrent antiretroviral therapy allowed provided regimen has been stable for at least 4 weeks
* No concurrent zidovudine
* No other concurrent KS-specific therapy
* No other concurrent investigational drugs, other than IND-approved antiretroviral agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-02; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Toxicity-related discontinuation rate | 28 days
Lytic induction rate | 28 days
Clinical response rate | 28 days
Accelerated KS progression rate | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Ambinder, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Mary Jo Lechowicz, MD, Study Chair — Georgia Cancer Center for Excellence at Grady Memorial Hospital
Locations (13):
- United States (13):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington